CLINICAL TRIAL: NCT03090594
Title: Diagnostic Performance and Complications of Transbronchial Cryobiopsy in Lung Transplant Patients According to the Number of Samples Obtained
Brief Title: Transbronchial Cryobiopsy in Lung Transplant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CB JKMT-2
Record Dates: First submitted 2017-03-14; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Lung Transplantation
Keywords: Cryoprobe; Bronchoscopy; Acute cellular rejection
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy (Other): Transbronchial biopsies with cryoprobe.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Is to obtain pulmonary parenchyma samples using a flexible bronchoscope.

SUMMARY:
Cryobiopsy has displaced the transbronchial biopsy (BTB) with forceps because it allows to obtain samples of more representative pulmonary parenchyma with more alveoli, less artifacts and a greater diagnostic yield. However, some authors report an increase in adverse effects such as hemorrhage and pneumothorax. The latest ISHLT (International Society for Heart and Lung Transplantation) consensus of 2007 recommends that with BTB with forceps a minimum of five tissue samples should be obtained that should contain more than 100 wells or the presence of two bronchioles to Which may be necessary between 3 and 17 samples. The optimal number of transbronchial cryobiopsies is unknown in order to obtain maximum performance with the lowest possible morbidity.

It is proposed to analyze the morphological and histopathological characteristics of each cryobiopsies individually and in order of extraction, to determine the sensitivity in the diagnosis of acute rejection as a function of the number of samples. Lung transplant patients, not admitted to critical units, with BTB indication will be included. A maximum of 6 samples will be obtained by flexible bronchoscope and under general anesthesia.

These data will allow to know the minimum number of specimens that guarantee a histological and / or bacteriological diagnosis of certainty with maximum effectiveness.

DETAILED DESCRIPTION:
Transbronchial biopsies (BPTB) will be performed using a flexible bronchoscope and the biopsy will be performed with cryoprobe (Erbokryo®). The patient undergoing the procedure will be intubated, sedated and relaxed under continuous monitoring (pulse oximetry, blood pressure, heart and respiratory rate), oxygen therapy with high flows and surveillance by anesthesiologist. The site where the biopsies will be performed will be determined based on an imaging study (chest x-ray and / or CT scan). The procedure will be performed according to the conventional technique, keeping the patient in apnea during the time that the cryobiopsies are taken to reduce the risk of pneumothorax. At most 6 samples will be obtained, and each one will be placed in an individual container listed in order of extraction. Bronchoalveolar lavage (3 aliquots of 30 mL sterile saline solution) will be performed in the same hemithorax. The samples obtained will be evaluated morphologically and sent to a microbiological and histopathological study, which will include a cell count. The data obtained will be coded.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary transplant patients with suspected rejection or infection requiring transbronchial biopsy

Exclusion Criteria:

* Respiratory failure refractory to oxygen therapy.
* Acute or subacute ischemic heart disease (last 4-6 weeks).
* Severe arrhythmias.
* Coagulation disorders: platelets <60,000-50,000 or Prothrombin time <60%.
* Lack of consent informed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-09-17 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of transbronchial biopsies with which a pathological diagnosis is obtained. The rejection graduation according to the criteria of the International Society for Heart Lung Transplantation (ISHLT). | 5-7 days.
  A maximum of 6 samples will be obtained.

SECONDARY OUTCOMES:
Number of alveoli, bronchi, bronchioles, blood vessels and pleura containing each biopsy. | 30 days.
  The Mese Software will be used. ¨Leica Application Suite X¨.
Number of complications related to the procedure. | 30 days.
  Complications related to the procedure: bleeding, pneumothorax, pneumonia, acute respiratory failure or need for hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Javier De Gracia, MD PhD, Principal Investigator — Respiratory department.; Karina Loor, MD, Study Chair — Respiratory department.; Mario Culebras, MD, Study Chair — Respiratory department.; Antonio Álvarez, MD, Study Chair — Respiratory department.
Locations (1):
- Hospital Vall de Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No